CLINICAL TRIAL: NCT01392053
Title: Assessment of the Effects of Massage Pain Relief in Nulliparous Women During the Active Phase of Labor
Brief Title: Massage for Pain Relief During the Active Phase of Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Silvana Maria Quintana, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FR259127
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Results first posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Pain
Keywords: labor; pain; massage
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Control Group (CG) that will receive the routine procedures of motherhood, but will be monitored and evaluated at the same time in the intervention group
- Massage Group (Experimental): Massage Group (GM):receive lumbosacral massage for 30 minutes, during uterine contractions between 4-5 cm of cervical dilation
  Interventions: Other: Lumbosacral Massage

INTERVENTIONS:
Other: Lumbosacral Massage — Massage Group (GM) will receive lumbosacral massage for 30 minutes, during uterine contractions between 4-5 cm of cervical dilation.
  Arms: Massage Group

SUMMARY:
The objective of this research is to evaluate the effect of massage therapy as a resource for pain relief during the active phase of labor. The research will be of type randomized controlled trial, consisting of low-risk nulliparous pregnant women admitted to the Referral Center for Women's Health in Ribeirão Preto. The mothers will be distributed in two groups (lumbosacral massage) and control (routine maternity) and will be assessed before and after therapy, which corresponds to 30 minutes between 4-5 cm of cervical dilation. The evaluation will be performed by numerical category scale, Diagram Location of Pain and Pain Questionnaire McGll (reduced form). After delivery will apply a customer satisfaction questionnaire.

DETAILED DESCRIPTION:
The pain in labor appears as a subjective experience, individual interaction involving a broad physiological, psychosocial and environmental influences, representing one of the main clinical signs of this phase. Despite presenting an important biological function, is today well established the need for their relief, since its persistence is associated with harmful effects on mother and fetus. Among the available non-pharmacological resources, we highlight the massage therapy that has shown positive effects in relieving pain and promoting the comfort of the mother. The objective of this research is to evaluate the effect of massage therapy as a resource for pain relief during the active phase of labor. The research will be of type randomized controlled trial, consisting of low-risk nulliparous pregnant women admitted to the Referral Center for Women's Health in Ribeirão Preto. The mothers will be distributed in two groups (lumbosacral massage) and control (routine maternity) and will be assessed before and after therapy, which corresponds to 30 minutes between 4-5 cm of cervical dilation. The evaluation will be performed by numerical category scale, Diagram Location of Pain and Pain Questionnaire McGll (reduced form). After delivery will apply a customer satisfaction questionnaire. After collecting the data, the groups are statistically analyzed using the linear regression model with mixed effects (fixed and random), taking into account a value of p <0.05 to obtain the statistical significance of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* literate
* A single fetus in vertex position
* Low-risk Pregnancy
* From 37 weeks of gestation
* Cervical dilatation from 4 cm with normal uterine dynamics in this phase
* Labor in early spontaneous
* No use of medications during the study period
* Absence of cognitive or psychiatric problems
* Intact membranes
* No risk factors associated
* You want to participate and signing the informed consent

Exclusion Criteria:

* Use of drugs or any procedure that aims to relieve pain
* Intolerance to the application of massage therapy
* Presence of dermatological conditions that indicate against the application of massage therapy

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Referral center for women's health Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Result] Chang MY, Wang SY, Chen CH. Effects of massage on pain and anxiety during labour: a randomized controlled trial in Taiwan. J Adv Nurs. 2002 Apr;38(1):68-73. doi: 10.1046/j.1365-2648.2002.02147.x. PMID 11895532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized and controlled non-inferiority clinical trial with a blind rater involving comparative analysis of a study group and a control group. The study included 46 parturients admitted to the Reference Center of Women's Health of Ribeirão Preto-MATER, state of São Paulo, Brazil, during the period from September 2009 to May 2010.
Pre-assignment Details: 149 women in labour were eligible, were excluded because their women 103 not attended the criteria for inclusion (primigesta, single fetus cephalic position, low-risk pregnancy, least 37 weeks, cervical dilation 4-5 cm, spontaneous onset of labor, no use of medication during the study period, intact membranes, and no associated with risk factors).
Period: Overall Study
Arm/Group | Control Group | Massage Group
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Massage Group | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 10 | 19
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19 (3.7) | 19 (3.2) | 19 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Massage Therapy in Pain Relief During Labor.
Description: The Visual Analogue Scale was used to assess the pain intensitiy after each procedure according to the study design. The VAS is a scale composed by a straight line printed on a paper measuring 100 milimeters, where only the 0 (Zero) and the 100 (one hundred) points are marked. The patient is then asked to mark this line accordingly to the intensity of the pain felt in that moment, considering 0 (Zero) to be no pain at all, and 100 (one hundred) to be the most unbearable pain ever suffered. The researcher would measure the distance, in milimeters, from the 0 (Zero)mm to the point were the patient marked, wich was considered to be the intensity of the pain felt by the patient in that moment. A reduction of 13mm or more in this scale is considered to be a significative pain reduction.
Time Frame: 30 minutes
Population: A pilot study was conducted previously to determine the size of the population needed. Using a paired sample t-test, with a power of 95% and 5% significance level, it was determined a minimum of 12 patients for Control Group and 16 patients for Massage Group
Measure: Mean (Standard Deviation); unit: milimeters
Arm/Group | Control Group | Massage Group
Number analyzed (Participants) | 23 | 23
milimeters
  Before Procedure | 68.7 (16.5) | 69.0 (14.5)
  After Procedure | 72.1 (15.4) | 51.7 (19.9)

2. Secondary Outcome: Pharmacological Analgesia Request According to the Cervical Dilation.
Description: In the institution where this study was conducted, the request for analgesia, made by the patient, is granted promptly. Considering that the further the cervyx dilation grows, the greater the pain intensity is, the cervical dilation was used as an indicator of the moment that the women in labour requested this procedure, and, therefore, could provide a comparison between methods.
Time Frame: 10 hours
Population: Of the 46 patients who where evaluated, only 1 (one) in each group didn't request pharmacological analgesia and, thus, were excluded of the analysis of this specific outcome
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Control Group | Massage Group
Number analyzed (Participants) | 22 | 22
centimeters | 6 (1.2) | 7 (1.3)

3. Secondary Outcome: Obstetric Outcomes - Delivery
Description: Labour can either occur via vaginal canal, also called natural birth, or via caesarian section, which is a surgical procedure used when either the mother or the baby are in distress.
Time Frame: 10 hours
Population: All patients of both groups were analyzed.
Measure: Number; unit: participants
Arm/Group | Control Group | Massage Group
Number analyzed (Participants) | 23 | 23
participants
  Vaginal | 19 | 17
  Caesarian section | 4 | 6

4. Secondary Outcome: Obstetric Outcomes - Duration of Labour
Description: The time elapsed between hospital admission and delivery was measured to compare the influence of the procedures established in the study design. It was defined two sets of measures dichotomizing the groups into "up to 7 hours" or "more than 7 hours".
Time Frame: 10 hours
Population: All patients in both groups were analyzed
Measure: Number; unit: percentage of participants
Arm/Group | Control Group | Massage Group
Number analyzed (Participants) | 23 | 23
percentage of participants
  Up to 7 hours | 83 | 57
  More than 7 hours | 17 | 43

5. Secondary Outcome: Obstetric Outcome - Moment of Corioamniorrhexis
Description: Corioamniorrhexis may occur during the normal evolution of labour or due to medical conditions. In this study, the moment when this event happened was associated to the dilation of the uterus cervyx, considering this to be a more reliable datum rather than the timelapse of labor. This outcome is measured in centimeter when the women is assessed by the doctor.
Time Frame: 10 hours
Population: All patients in both groups were analyzed
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Control Group | Massage Group
Number analyzed (Participants) | 23 | 23
centimeters | 8.0 (1.7) | 7.5 (1.7)

6. Secondary Outcome: Obstetric Outcomes - Moment of Utilization of Oxytocin
Description: Oxytocin is a drug used to induce or enhance the muscular activity of the uterus. In this study, the moment when this event happened was associated to the dilation of the uterus cervyx, considering this to be a more reliable data rather than the timelapse of labor. This outcome is measured in centimeter when the women is assessed by the doctor.
Time Frame: 10 hours
Population: All patients in both groups were analyzed
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Control Group | Massage Group
Number analyzed (Participants) | 23 | 23
centimeters | 6.0 (2.0) | 5.0 (2.8)

7. Secondary Outcome: Satisfaction of Mothers With the Presence of a Professional by Their Side During the Study Period.
Description: Considering the first labour to be a unique experience to every women, and also a moment of many doubts and insecurities, it is considered that the presence of a healthcare professional, providing information and support, during this moment, could be benefitial to most first time mothers. Therefore, the presence of a physiotherapist could have helped minimize the suffering in both groups. The questionnaire applied after labour intended to assess how most women felt regarding this subject.
Time Frame: 30 minutes
Population: All patients participatin in the study answered a satisfaction questionnaire after labour.
Measure: Number; unit: participants
Arm/Group | Control Group | Massage Group
Number analyzed (Participants) | 23 | 23
participants
  Considered important presence of physiotherapist | 23 | 23
  Rated excellent the therapy received | 16 | 15

ADVERSE EVENTS:
Arm/Group | Control Group | Massage Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The influence of the pain of other women in labor or under the effect of childbirth analgesia; Accompanying with no physical or emotional preparation; Brazilian culture, which associates pain with suffering.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No